CLINICAL TRIAL: NCT05123326
Title: Prospective Evaluation of Coagulation Status and Thromboelastometry Guided Management of Genetic and Acquired Thrombophilia in Patients With Portal Vein Thrombosis and Budd-Chiari Syndrome
Brief Title: Global Coagulation Assessment in Portal Vein Thrombosis and Budd-Chiari Syndrome
Acronym: Liv-Thrombus
Status: Recruiting | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: PGI/IEC/2021/001451
Record Dates: First submitted 2021-11-03; First posted 2021-11-17 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hepatic Vein Thromboses; Hepatic Venous Outflow Obstruction; Portal Vein Thrombosis; Portal Hypertension, Noncirrhotic; Portal Vein Occlusion; Portal Vein Embolism; JAK2 Mutation; CALR Gene Mutation; Prothrombin G20210A; Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Budd-Chiari Syndrome; Hypertension, Portal; Hemostatic Disorders | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and serum samples for thrombophilia evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PVT: Portal Vein Thrombosis (PVT) refers to partial or complete occlusion of the portal vein lumen by a blood clot or its replacement by multiple collateral vessels with the hepato-petal flow, commonly known as 'portal cavernoma.' 240 patients to be recruited
  Interventions: Diagnostic Test: Rotational thromboelastometry; Diagnostic Test: Genetic tests for Thrombophilia; Diagnostic Test: ELISA tests/ Functional assays
- HVOTO: Occlusion of two or more hepatic veins. 100 patients
  Interventions: Diagnostic Test: Rotational thromboelastometry; Diagnostic Test: Genetic tests for Thrombophilia; Diagnostic Test: ELISA tests/ Functional assays

INTERVENTIONS:
Diagnostic Test: Rotational thromboelastometry — ROTEM/ Sonoclot tests will be done in all patients at enrolment and after initiating anticoagulation in those who are eligible for the same.
  Other Names: Global coagulation test
Diagnostic Test: Genetic tests for Thrombophilia — Tests for JAK2 mutation, CAL R mutation and Factor V Leiden mutation will be done.
Diagnostic Test: ELISA tests/ Functional assays — Antithrombin III, Protein C, Protein S, Factor VIII, VWF using commercial assays

SUMMARY:
Portal vein thrombosis is defined as partial or complete occlusion of the portal vein lumen by the blood clot or its replacement by multiple collateral vessels with the hepato-petal flow, known as 'portal cavernoma'. [1,2] Based on the published literature, 15-25% of patients with cirrhosis have portal vein thrombosis (PVT) [3], and 35-50% of patients with hepatocellular carcinoma (HCC) have malignant PVT [4] compared to 1-3.8 per 100,000 patients in the general population. [5] The reported cumulative incidence of PVT in patients of Child-Pugh A and B is 4.6% and 10.7% at 1 and 5 years respectively with higher incidence among those with decompensated disease or with an underlying hypercoagulable disorder. [6]. Similarly, the prevalence of PVT in compensated cirrhosis is around 1% which increases to 8 - 25% in liver transplant (LT) candidates and 40% in patients with hepatocellular carcinoma (HCC) [7,8]. Based on the published literature 7-9 % of all chronic liver disease patients have hepatic vein outflow tract obstruction (HVOTO) in the Indian population. [9] HVOTO is defined as obstruction to hepatic venous outflow at any site from the right atrium inlet to the small hepatic venules. The Budd-Chiari syndrome (BCS) results from occlusion of one or more hepatic veins (HV) and/or the inferior vena cava (IVC). In the West, the most common cause is HV occlusion by thrombosis. More recent Indian studies have however shown that isolated HV and combined IVC+HV obstruction are now more common. [10]

In the post COVID-19 era, there has been great interest in the prothrombotic states associated with the SARS-Cov-2 virus infection, and the adverse effects of some vaccines. [11] With the availability of better molecular tests for hypercoagulable states, use of global coagulation tests (GCT) like rotational thromboelastometry (ROTEM), thromboelastography (TEG) and Sonoclot, use of therapeutic procedures like Transjugular intrahepatic portosystemic shunt (TIPS), availability of novel oral anticoagulants (NOAC), the natural course of disease can be changed with good outcomes. [12] Standard Coagulation tests (SCTs) like PT, aPTT, and platelet count are not predictive of bleeding or coagulation risk as they exclude the cellular elements of hemostasis and are unable to assess the effect of thrombomodulin and cannot assess the stage of the coagulation pathway which is affected. Global coagulation tests provide dynamic information on the coagulation pathway that is not available from conventional tests. [13]

DETAILED DESCRIPTION:
Our proposed study is important for the following 4 reasons.

1. SCTs cannot be used to demonstrate the thrombomodulin mediated normal thrombin generation in patients with liver disease, so the monitoring of such patient using global coagulation tests can be validated. The use of point-of-care global coagulation tests like ROTEM and Sonoclot enables us to identify the true prothrombotic and hypocoagulable states which can be used to assess for increased clot strength, clot formation time, and indicate hyperfibrinolysis. The use of conventional tests like prothrombin time, partial thromboplastin time and INR cannot bolster the therapeutic strategy.
2. This study will also help to determine role of global coagulation tests rather than PT/INR /aPTT in monitoring the dose and response of anticoagulants like vitamin K antagonists and novel oral anticoagulants (NOAC) in patients who are on therapeutic anticoagulation for HVOTO/PVT.
3. This study will also help to determine the prevalence and role of CALR, JAK2V617F, factor V Leiden mutations in patients with PVT and HVOTO in our population.
4. We will also be prospectively assessing the rate of thrombophilia complications in the Post COVID-19 era, and the study will generate information regarding new incidence of PVT/HVOTO in those exposed to COVID-19.

Therefore, the current study is the need of the hour, as we intend to assess the relevance of PVT and outcomes, test the genetic predisposition of Indian patients to hyper coagulable states, develop anticoagulation algorithms using NOAC, and determine the true burden on disease in India.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Either gender
* Age:18 - 65 years of age
* Patient with portal vein thrombosis documented on imaging (USG with color doppler, CECT abdomen and CEMRI abdomen

Exclusion Criteria:

* Patients who do not consent to the study.
* Patient with pregnancy and lactation
* Patients with a history of blood transfusions in the last two weeks
* Patients who are too sick to undergo screening tests.
* Patients on hemodialysis
* Chronic heart failure and chronic pulmonary or end-stage renal disease
* Patients who are on plasma therapy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with PVT and HVOTO fitting the inclusion criteria will be prospectively enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Clinical presentation | At enrolment
  Number of participants with clinical and imaging evidence of PVT and HVOTO in our patient population
Clinical presentation- Extent of disease | At enrolment
  Grading of PVT and HVOTO in our patient population
Occurrence of new thrombotic complications | At enrolment-3 years
  Description of new sites of thrombosis spectrum of PVT and HVOTO in our patient population
Occurrence of all thrombotic complications after anticoagulation | At enrolment-3 years
  Description of new sites of thrombosis spectrum of PVT and HVOTO after anticoagulation
Comparison of performance of standard coagulation tests vs. global coagulation tests to determine the hypercoagulable defect | At enrolment
  PT aPTT INR
Comparison of performance of global coagulation tests to determine the hypercoagulable defect | At enrolment
  ROTEM/Sonoclot

SECONDARY OUTCOMES:
Assessment of genetic predisposition of hypercoagulable states in PVT and HVOTO | At enrolment
  JAK2, CALR, Factor V Leiden mutation
Assessment of genetic predisposition of hypercoagulable states in PVT and HVOTO | At enrolment
  CALR mutation test
Assessment of genetic predisposition of hypercoagulable states in PVT and HVOTO | At enrolment
  Factor V Leiden mutation
Assessment of genetic predisposition of hypercoagulable states in PVT and HVOTO | At enrolment
  JAK2 mutation test
Occurrence of new hemorrhagic complications | At enrolment-3 years
  Sites of bleeding in patients who are not on anticoagulation
Occurrence of new hemorrhagic complications in anticoagulated patients | At enrolment-3 years
  Sites of bleeding in patients who are on anticoagulation

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, MD DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Choose Any State/Province, India

IPD SHARING:
Plan to Share IPD: Undecided